CLINICAL TRIAL: NCT05165641
Title: Segmental Spinal Anesthesia for Small-incision Cholecystectomy in a Field Hospital
Acronym: SPICHOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avicenna Military Hospital (Other)
Responsible Party: Principal Investigator, Younes Aissaoui, MD, Professor of anesthesia and intensive care medicine, Avicenna Military Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPICHOL AvicennaMH
Record Dates: First submitted 2017-08-10; First posted 2021-12-21 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Gall Stones (& [Calculus - Gall Bladder]); Anesthesia
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- segmental spinal anesthesia (Other): thoracic spinal anesthesia at T 10 level
  Interventions: Procedure: segmental spinal anesthesia

INTERVENTIONS:
Procedure: segmental spinal anesthesia — Spinal anesthesia was performed at a lower thoracic level with the patient in the sitting position. After local anesthesia with 1% lidocaine, the spinal puncture was done in the 10th thoracic intervertebral space (T 10) through a median approach. A 27 Gg pencil-point needle with an introducer was used (marquee). To identify T 10, the vertebra prominens (C7) was palpated and the spinous processes were palpated caudally [ref}. Two senior anesthesiologists performed all the spinal punctures. The progression of the spinal needle was cautious and soft. The effort was made to stop the needle progression just after the tactile perception of the dura mater. Once the flow of cerebrospinal fluid was obtained, 1.5 ml of hyperbaric bupivacaine 5mg/ml (=7.5 mg) mixed with 0.5 ml of fentanyl 50 µg/ml (= 25 µg) was injected and the spinal needle removed.

SUMMARY:
Providing safe and efficient anesthesia and in a field hospital is a challenging situation. This study investigated the feasibility and safety of thoracic spinal anesthesia for small-incision open cholecystectomy in a deployed field hospital.

DETAILED DESCRIPTION:
This study was conducted in a field hospital deployed in a rural area of the middle Atlas in Morocco during the winters of 2016 and 2017. The Middle Atlas is a part of the Atlas mountain range which is usually blocked and isolated by snow during the winter. The hospital deployed was an inflatable tent hospital self-contained and self-sufficient. This field hospital included the following components: a patient's ward (sixty beds), an operating theater with one surgical table, a recovery room with 2 beds, a laboratory, an X-ray unit, a pharmacy, and several exams rooms.

After approval by the Ethical review board of Avicenna Military Hospital, Marrakech, Morocco (CERB7/2016), written informed consent was obtained from patients who agreed to participate in the study.

The inclusion criteria were: uncomplicated symptomatic cholelithiasis confirmed by preoperative ultrasound, age 18 years or older and American society of anesthesiologists (ASA) physical status I, II or III. Exclusion criteria were: patients with acute cholecystitis, suspected common bile duct stones, previous abdominal surgery, bleeding diathesis, spinal abnormality, and allergy to any drug used in the study.

Patients were interviewed and examined by an anesthesiologist in a preoperative visit several days before surgery. On arrival in the operating room the patient's non-invasive blood pressure, oxygen saturation, and heart rate were monitored. Heart rate and blood pressure were recorded every five minutes. Intravenous access was established in the forearm with an 18 Gauge catheter and patients received a preload with 10 ml/Kg of normal saline. Patients were given 1mg midazolam intravenously for anxiolysis and oxygen 2-3 l /min was administered by a nasal cannula. Cefazolin 2 g was injected as antimicrobial prophylaxis. Antiemetic prophylaxis was also carried out with dexamethasone 4 mg IV.

Spinal anesthesia was performed at a lower thoracic level with the patient in the sitting position. After local anesthesia with 1% lidocaine, the spinal puncture was done in the 10th thoracic intervertebral space (T 10) through a median approach. A 27 Gg pencil-point needle with an introducer was used (marquee). To identify T 10, the vertebra prominens (C7) was palpated and the spinous processes were palpated caudally. Two senior anesthesiologists performed all the spinal punctures. The progression of the spinal needle was cautious and soft. The effort was made to stop the needle progression just after the tactile perception of the dura mater. Once the flow of cerebrospinal fluid was obtained, 1.5 ml of hyperbaric bupivacaine 5mg/ml (=7.5 mg) mixed with 0.5 ml of fentanyl 50 µg/ml (= 25 µg) was injected and the spinal needle removed. Patients were asked to report any pain or paresthesia during the puncture. The patient was then placed in a supine horizontal position. The level of sensory block was assessed every 2 minutes (pinprick method). After an adequate sensory block was obtained (T4 - T 12), surgery was allowed to start. The nasogastric tube was not inserted unless the surgeon required it.

Patients were invited to report any discomfort or pain during surgery. Patients were asked to assess any eventual pain on a numeric rating scale ranging from 0 (no pain) to 10 (worst possible pain). Perioperative pain scores were collected at skin incision and perioperative pain and anxiety were treated with boluses of fentanyl 50 µg (maximum 100 µg) and midazolam 1 mg (maximum 5 mg). The need for additional sedation/analgesia and the doses administered were recorded. Patients were informed about the possibility of switching to general anesthesia (GA). Criteria for conversion to GA were: failure of spinal anesthesia, pain score > 4 despite a maximum dose of fentanyl, and difficult surgical conditions.

Two experienced surgeons performed all operations. Small incision open cholecystectomy was performed with a 6 to 8 cm long transverse incision over the right rectus abdominis muscle, as described by Rosenmuller [ref]. Surgeon s satisfaction was evaluated by asking surgeons to assess the operative conditions on a numeric scale of 0 to 10 (0: worst surgical conditions, 10: best operative conditions). At the time of skin closure, a wound infiltration (muscular compartment and subcutaneous fat) with 15 to 20ml of bupivacaine 0.25% was made.

The duration of surgery and perioperative incidents (hypotension, bradycardia nausea, and/or vomiting) were recorded. Hypotension defined as a drop in the mean arterial blood pressure (MAP) ≥20% below baseline was managed by IV boluses of ephedrine 6 mg. Bradycardia was defined as heart rate <50 and treated with atropine 0.50 mg. Post-operative events were also recorded: nausea and vomiting, urinary retention, pruritus, headache, or neurologic symptom. Patients were discharged the day after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated symptomatic cholelithiasis
* American society of anesthesiologists (ASA) physical status I, II, or III

Exclusion Criteria:

* patients with acute cholecystitis
* suspected common bile duct stones
* previous abdominal surgery
* bleeding diathesis
* spinal abnormality
* allergy to any drug used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of segmental spinal anesthesia for small-incision open cholecystectomy in a field hospital | intraoperatively
  Patients' peroperative pain scores assessed on a numeric rating scale ranging from 0 (no pain) to 10 (worst possible pain)
Hemodynamic tolerance of segmental spinal anesthesia. | intraoperatively
  Heart rate (beats per minute): monitored and recorded every 5 minutes:
Hemodynamic tolerance of segmental spinal anesthesia. | intraoperatively
  Non-invasive blood pressure (mmHg): monitored and recorded every 5 minutes:
Respiratory safety of segmental spinal anesthesia. | intraoperatively
  Respiratory rate (breaths per minute): monitored and recorded every 5 minutes.
Respiratory safety of segmental spinal anesthesia. | intraoperatively
  Pulse oximetry (%): monitored and recorded every 5 minutes.

SECONDARY OUTCOMES:
surgeon's satisfaction with anesthesia technique | intraoperatively
  numeric scale from 0 to 10 (0: worst surgical conditions, 10: best operative conditions)
patient satisfaction with anesthesia technique | 24 hours postoperatively
  numeric rating scale from 0 to 10
postoperative adverse effects | 24 hours postoperatively
  nausea and vomiting, urinary retention, pruritus, headache, neurologic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Younes Aissaoui, Principal Investigator — Avicenna Military Hospital

IPD SHARING:
Plan to Share IPD: No